CLINICAL TRIAL: NCT05011331
Title: The Effect of a Custom Pillow on Sleep Quality in Patients With Nonoperative Rotator Cuff Syndrome: a Prospective Randomized Study
Brief Title: The Effect of a Custom Pillow on Sleep Quality in Patients With Nonoperative Rotator Cuff Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Amenity Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1620695
Record Dates: First submitted 2021-08-02; First posted 2021-08-18 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MedCline Shoulder Relief System (Experimental): Patients who will receive the MedCline Shoulder Relief System pillow
  Interventions: Device: MedCline Shoulder Relief System
- Control (Active Comparator): Patients who will not receive the MedCline Shoulder Relief System pillow
  Interventions: Device: MedCline Shoulder Relief System

INTERVENTIONS:
Device: MedCline Shoulder Relief System — Patients will receive a customized pillow to aid with sleep

SUMMARY:
The objective of this study is to determine if a pillow sleep aid improves sleep quality in the short term for patients who have shoulder pain from a rotator cuff injury and are being managed non-operatively.

DETAILED DESCRIPTION:
Patients who have shoulder pain from a rotator cuff injury will be identified in the outpatient clinic and offered the chance to enroll in the study. Informed consent will be obtained. There will be two groups of patients in this study; those that receive the pillow sleep aid (the intervention group) and those that do not (the control group). The pillow sleep aid that will be investigated in this project is the "MedCline Shoulder Relief System," a product of Amenity Health Inc.. The pillow will be delivered to the intervention group at no cost. Patients in both groups will be prescribed the same physical therapy protocols. At the end of the trial period, patients in the control group will be offered the option to receive a pillow. Those that accept will be surveyed at similar intervals as the original intervention group.

ELIGIBILITY:
Inclusion Criteria:

* age >18 and a diagnosis of rotator cuff syndrome which is being treated non-operatively.

Exclusion Criteria:

* history of prior shoulder surgery, receiving a corticosteroid injection at initial visit, lack of mailing address, non-English speaking patient, inability to sleep on one's side, preexisting clinical insomnia and obstructive sleep apnea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-10-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Sleep Difficulty as Assessed as Assessed Using the Insomnia Severity Index (ISI) | Baseline, two weeks, six weeks
  The ISI assesses sleep difficulty using a 5 point Likert Scale, where a lower score is better
Change from Baseline in Pain Scores on the Visual Analog Scale (VAS) | Baseline, two weeks, six weeks
  The VAS utilizes a scale from 0-10 where a high score indicates more pain
Change in Quality of Life as Assessed Using the Euroqol (EQ-5D) | Baseline, two weeks, six weeks
  The EQ-5D assesses quality of life with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
Change in Shoulder Function as Assessed Using the American Shoulder and Elbow Surgeons Shoulder Score (ASES) | Baseline, two weeks, six weeks
  The ASES is a 100-point scale that consists of two dimensions: pain and activities of daily living. There is a pain scale worth 50 points and ten activities of daily living questions worth 50 points
Change in Shoulder Function as Assessed Using the Single Assessment Numeric Evaluation (SANE) | Baseline, two weeks, six weeks
  SANE assesses shoulder function via 1 question as a percentage of normal (0-100 scale with 100 being normal)
Change in Shoulder Function as Assessed Using the Western Ontario Rotator Cuff Index (WORC) | Baseline, two weeks, six weeks
  WORC utilizes 21 questions where each question uses a visual analog scale, a line with a 0-100 scale where 0 represents no difficulty. It asks about shoulder pain in 5 different domains, physical symptoms, sports, work, social, and emotions

CONTACTS AND LOCATIONS:
Overall Officials: E S Paxton, MD, Principal Investigator — University Orthopedics
Locations (1):
- University Orthopedics, East Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No